CLINICAL TRIAL: NCT04631562
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Single and Multiple Ascending Dose Study of Subcutaneous and Intravenous ALXN1820 in Healthy Participants
Brief Title: Study of ALXN1820 in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: ALXN1820-HV-101; 2021-002472-39 (EudraCT Number)
Record Dates: First submitted 2020-11-13; First posted 2020-11-17 (Actual); Results first posted 2024-03-15 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-07

CONDITIONS: Healthy
Keywords: ALXN1820; Properdin; Pharmacodynamics; Pharmacokinetics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ALXN1820 (Experimental): Participants will receive ALXN1820 SC or ALXN1820 IV according to their assigned cohort. ALXN1820 SC will be evaluated in single and multiple ascending doses while ALXN1820 IV will be evaluated in a single dose cohort only.
  Interventions: Drug: ALXN1820 SC; Drug: ALXN1820 IV
- Placebo (Placebo Comparator): Participants will receive Placebo SC or Placebo IV according to their assigned cohort.
  Interventions: Drug: Placebo SC; Drug: Placebo IV

INTERVENTIONS:
Drug: ALXN1820 SC — ALXN1820 SC will be administered as a manual SC push or SC infusion via a syringe pump. Doses will range from 12.5 milligrams (mg) to a maximum of 2250 mg. Multiple dosing duration will range from 3 to 5 weeks.
  Arms: ALXN1820
Drug: ALXN1820 IV — ALXN1820 IV (450 mg) will be administered as an IV infusion.
  Arms: ALXN1820
Drug: Placebo SC — Placebo SC will be administered as a manual SC push or SC infusion via a syringe pump.
  Arms: Placebo
Drug: Placebo IV — Placebo IV will be administered as an IV infusion.
  Arms: Placebo

SUMMARY:
This is a Phase 1, randomized, double-blind, placebo-controlled single and multiple ascending dose study designed to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, and immunogenicity of ALXN1820 administered subcutaneously (SC) (ALXN1820 SC) and intravenously (IV) (ALXN1820 IV).

DETAILED DESCRIPTION:
This study will include up to 10 different dosing cohorts, with each cohort consisting of 2 groups (ALXN1820 group, placebo group). Participants will be randomly assigned in a 3:1 ratio to each of these 2 groups, respectively, within all 10 cohorts, to receive either a single or multiple doses of ALXN1820 SC, a single dose of ALXN1820 IV, or a single or multiple doses of placebo.

The study will be conducted in healthy adult participants and will also include a multiple SC dose cohort in healthy participants of Japanese descent.

ELIGIBILITY:
Inclusion Criteria:

* Body weight 50 to 100 kilograms (kg); body mass index 17 to 32 kg/meter squared.
* Cohort 9 only: Japanese participants (defined as those participants whose parents and grandparents are both Japanese and who have spent less than 5 years outside of Japan).
* Satisfactory medical assessment.
* Must follow protocol-specified contraception guidance while on treatment and for up to 6 months after last dose.
* Vaccination requirement:

  * Vaccination with tetravalent meningococcal conjugate vaccine at least 56 days and not more than 2 years, 6 months prior to dosing;
  * Vaccination with serogroup B meningococcal vaccine at least 56 days prior to dosing, with a booster at least 28 days prior to dosing, with at least 28 days between the first and second injections.

Exclusion Criteria:

* Current/recurrent diseases or relevant medical history.
* History of any Neisseria infection.
* Hepatitis B/C, human immunodeficiency virus.
* History of latent or active tuberculosis (TB), or positive TB test.
* Active systemic infection within 14 days of dosing.
* Risk of meningococcal infections due to living/working conditions.
* History of complement deficiency or complement activity below the reference range.
* Participation in a clinical study within 90 days or 5 half lives of the investigational agent (whichever is longer) before initiation of dosing on Day 1.
* Participation in more than 1 clinical study of a monoclonal antibody (mAb), or participation in a clinical study of a mAb within the 6 months or 5 half lives of the mAb (whichever is longer) prior to screening.
* Acquired complement deficiencies (for example, those receiving eculizumab).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2021-01-13 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Research Site, Herston, Australia
- Research Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sandhu A, Shen T, Herrero PM, Yuan CX, Qureshi S, Jiang X, Sheng Y, Gasteyger C, Dai Y. Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Immunogenicity of ALXN1820 (Tarperprumig) in Healthy Adults: Results of a Phase I Study. Clin Transl Sci. 2025 Apr;18(4):e70190. doi: 10.1111/cts.70190. PMID 40134111

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: ALXN1820 12.5 mg SC: Healthy participants received a single dose of ALXN1820 12.5 mg subcutaneous (SC) injection on Day 1.
- Cohort 2: ALXN1820 50 mg SC: Healthy participants received a single dose of ALXN1820 50 mg SC injection on Day 1.
- Cohort 3: ALXN1820 150 mg SC: Healthy participants received a single dose of ALXN1820 150 mg SC injection on Day 1.
- Cohort 4: ALXN1820 450 mg SC: Healthy participants received a single dose of ALXN1820 450 mg SC injection on Day 1.
- Cohort 5: ALXN1820 450 mg IV: Healthy participants received a single dose of ALXN1820 450 mg intravenous (IV) infusion on Day 1.
- Cohort 6: ALXN1820 1200 mg SC: Healthy participants received a single dose of ALXN1820 1200 mg SC injection on Day 1.
- Cohort 8: ALXN1820 150 mg SC (QW*5): Healthy participants received multiple doses of ALXN1820 150 mg SC injection once weekly (QW) for 5 weeks.
- Cohort 9: ALXN1820 150 mg SC (QW*5): Healthy Japanese participants received multiple doses of ALXN1820 150 mg SC injection once weekly for 5 weeks.
- All Placebo: Healthy participants received placebo matched to ALXN1820 SC injection or IV infusion.
Period: Overall Study
Arm/Group | Cohort 1: ALXN1820 12.5 mg SC | Cohort 2: ALXN1820 50 mg SC | Cohort 3: ALXN1820 150 mg SC | Cohort 4: ALXN1820 450 mg SC | Cohort 5: ALXN1820 450 mg IV | Cohort 6: ALXN1820 1200 mg SC | Cohort 8: ALXN1820 150 mg SC (QW*5) | Cohort 9: ALXN1820 150 mg SC (QW*5) | All Placebo
Started | 5 | 6 | 5 | 5 | 5 | 6 | 7 | 6 | 15
Received at Least 1 Dose of Study Drug | 5 | 6 | 5 | 5 | 5 | 6 | 7 | 6 | 15
Completed | 5 | 6 | 5 | 4 | 5 | 6 | 6 | 5 | 14
Not Completed | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Set included all participants who received at least 1 dose of study drug.
Groups:
- Cohort 1: ALXN1820 12.5 mg SC: Healthy participants received a single dose of ALXN1820 12.5 mg SC injection on Day 1.
- Cohort 5: ALXN1820 450 mg IV: Healthy participants received a single dose of ALXN1820 450 mg IV infusion on Day 1.
- Cohort 8: ALXN1820 150 mg SC (QW*5): Healthy participants received multiple doses of ALXN1820 150 mg SC injection once weekly for 5 weeks.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: ALXN1820 12.5 mg SC | Cohort 2: ALXN1820 50 mg SC | Cohort 3: ALXN1820 150 mg SC | Cohort 4: ALXN1820 450 mg SC | Cohort 5: ALXN1820 450 mg IV | Cohort 6: ALXN1820 1200 mg SC | Cohort 8: ALXN1820 150 mg SC (QW*5) | Cohort 9: ALXN1820 150 mg SC (QW*5) | All Placebo | Total
Number analyzed (Participants) | 5 | 6 | 5 | 5 | 5 | 6 | 7 | 6 | 15 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 6 | 5 | 5 | 5 | 6 | 7 | 6 | 15 | 60
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 1 | 3 | 2 | 3 | 5 | 0 | 9 | 32
  Male | 2 | 0 | 4 | 2 | 3 | 3 | 2 | 6 | 6 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
  Not Hispanic or Latino | 5 | 4 | 5 | 4 | 3 | 6 | 7 | 6 | 12 | 52
  Unknown or Not Reported | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 6 | 3 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  White | 3 | 5 | 4 | 3 | 5 | 5 | 7 | 0 | 11 | 43
  More than one race | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-related Adverse Events (TEAEs) For ALXN1820 SC And ALXN1820 IV
Description: An adverse event (AE) was defined as any unfavorable and unintended sign (for example, including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product or procedure, whether or not considered related to the medicinal product or procedure, which occurred during the course of the clinical study. TEAEs were defined as any AEs that commenced after the start of administration of study intervention. Serious AEs (SAEs) were defined as any untoward medical occurrence that met at least 1 of the following serious criteria: resulted in death, was life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, other medically important serious event. A summary of all SAEs and Other AEs (nonserious) regardless of causality is located in the 'Reported AEs' Section.
Time Frame: Cohorts 1 to 6: Baseline up to Day 127; Cohorts 8 to 9: Baseline up to Day 155
Population: The Safety Set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: ALXN1820 12.5 mg SC | Cohort 2: ALXN1820 50 mg SC | Cohort 3: ALXN1820 150 mg SC | Cohort 4: ALXN1820 450 mg SC | Cohort 5: ALXN1820 450 mg IV | Cohort 6: ALXN1820 1200 mg SC | Cohort 8: ALXN1820 150 mg SC (QW*5) | Cohort 9: ALXN1820 150 mg SC (QW*5) | All Placebo
Number analyzed (Participants) | 5 | 6 | 5 | 5 | 5 | 6 | 7 | 6 | 15
Participants | 1 | 0 | 0 | 4 | 2 | 0 | 1 | 3 | 2

2. Secondary Outcome: Area Under The Concentration-time Curve (AUC) From Time 0 (Dosing) To Time Infinity (AUC0-inf) And AUC During The Dosing Interval (AUCtau) of Serum ALXN1820 For Single Dose Cohorts
Time Frame: Up to 126 days following the first day of dosing
Population: The Pharmacokinetic (PK) Set included all participants who received at least 1 dose of study drug and had at least 1 post-dose PK concentration measured. As per pre-specified analysis, only data for Cohorts 1-6 were collected for this Outcome Measure. Here, number analyzed (n) signifies those participants who were evaluable at specified categories.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*micrograms/milliliters
Arm/Group | Cohort 1: ALXN1820 12.5 mg SC | Cohort 2: ALXN1820 50 mg SC | Cohort 3: ALXN1820 150 mg SC | Cohort 4: ALXN1820 450 mg SC | Cohort 5: ALXN1820 450 mg IV | Cohort 6: ALXN1820 1200 mg SC
Number analyzed (Participants) | 5 | 6 | 5 | 5 | 5 | 6
hours*micrograms/milliliters
  AUC0-inf: number analyzed (Participants) | 1 | 6 | 5 | 4 | 5 | 6
  AUC0-inf | 1708.745740 (NA) — NA signifies that geometric coefficient of variation was not evaluable as there was only 1 participant. | 11871.887397 (18.11) | 22447.444516 (24.22) | 65994.232565 (23.56) | 70222.568018 (13.41) | 157445.098602 (15.80)
  AUCtau | 1301.090561 (35.33) | 11356.654811 (18.25) | 21767.138401 (24.61) | 56467.567738 (37.45) | 69126.480691 (13.16) | 151825.555391 (15.02)

3. Secondary Outcome: Area Under The Concentration-time Curve During The Dosing Interval (AUCtau) Of Serum ALXN1820 For Multiple Dose Cohorts
Time Frame: Up to 154 days following the first day of dosing
Population: The Pharmacokinetic Set included all participants who received at least 1 dose of study drug and had at least 1 post-dose PK concentration measured. Here, Number of participants analyzed signifies those who were evaluable for this outcome measure. As per pre-specified analysis, only data for Cohorts 8 and 9 were collected for this Outcome Measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*micrograms/milliliters
Arm/Group | Cohort 8: ALXN1820 150 mg SC (QW*5) | Cohort 9: ALXN1820 150 mg SC (QW*5)
Number analyzed (Participants) | 6 | 5
hours*micrograms/milliliters | 13047.247486 (11.96) | 14895.697459 (6.63)

4. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) Of Serum ALXN1820 For Single Dose Cohorts
Time Frame: Up to 126 days following the first day of dosing
Population: The Pharmacokinetic Set included all participants who received at least 1 dose of study drug and had at least 1 post-dose PK concentration measured. As per pre-specified analysis, only data for Cohorts 1-6 were collected for this Outcome Measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms/milliliters
Arm/Group | Cohort 1: ALXN1820 12.5 mg SC | Cohort 2: ALXN1820 50 mg SC | Cohort 3: ALXN1820 150 mg SC | Cohort 4: ALXN1820 450 mg SC | Cohort 5: ALXN1820 450 mg IV | Cohort 6: ALXN1820 1200 mg SC
Number analyzed (Participants) | 5 | 6 | 5 | 5 | 5 | 6
micrograms/milliliters | 2.346 (17.85) | 12.892 (10.48) | 29.342 (22.53) | 99.256 (33.98) | 162.518 (46.73) | 246.140 (17.14)

5. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) Of Serum ALXN1820 For Multiple Dose Cohorts
Time Frame: Up to 154 days following the first day of dosing
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms/milliliters
Arm/Group | Cohort 8: ALXN1820 150 mg SC (QW*5) | Cohort 9: ALXN1820 150 mg SC (QW*5)
Number analyzed (Participants) | 6 | 5
micrograms/milliliters | 90.53 (12.40) | 100.97 (7.94)

6. Secondary Outcome: Change From Baseline in Serum Concentrations Of Total Properdin For ALXN1820 SC And ALXN1820 IV-Single Dose Cohorts
Time Frame: Baseline, Day 127
Population: The Pharmacodynamic Set included all participants who received at least 1 dose of study drug and had evaluable properdin concentration, CAP or complement classical pathway activity data. Here, Number of participants analyzed signifies those who were evaluable for this outcome measure. As per pre-specified analysis, only data for Cohorts 1-6 and the placebo arm were collected for this Outcome Measure.
Measure: Mean (Standard Deviation); unit: micrograms/milliliters
Groups:
- Placebo: Non-Japanese participants received placebo matched to ALXN1820 SC injection or IV infusion.
Arm/Group | Cohort 1: ALXN1820 12.5 mg SC | Cohort 2: ALXN1820 50 mg SC | Cohort 3: ALXN1820 150 mg SC | Cohort 4: ALXN1820 450 mg SC | Cohort 5: ALXN1820 450 mg IV | Cohort 6: ALXN1820 1200 mg SC | Placebo
Number analyzed (Participants) | 5 | 6 | 5 | 5 | 5 | 6 | 11
micrograms/milliliters | 3.744 (0.8941) | 2.093 (1.3870) | 1.788 (1.7589) | 5.580 (3.1652) | 3.014 (2.0181) | 15.017 (7.1687) | 1.240 (1.4712)

7. Secondary Outcome: Change From Baseline in Serum Concentrations Of Free Properdin For ALXN1820 SC And ALXN1820 IV-Single Dose Cohorts
Time Frame: Baseline, Day 127
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: nanograms/milliliters
Arm/Group | Cohort 1: ALXN1820 12.5 mg SC | Cohort 2: ALXN1820 50 mg SC | Cohort 3: ALXN1820 150 mg SC | Cohort 4: ALXN1820 450 mg SC | Cohort 5: ALXN1820 450 mg IV | Cohort 6: ALXN1820 1200 mg SC | Placebo
Number analyzed (Participants) | 5 | 6 | 5 | 5 | 5 | 6 | 11
nanograms/milliliters | 848.0 (508.40) | 1096.7 (1815.02) | 1200.0 (1078.61) | 20.8 (2667.17) | 1188.4 (975.93) | 5171.8 (910.95) | -26.6 (1749.15)

8. Secondary Outcome: Change From Baseline In Serum Concentrations of Total Properdin For ALXN1820 SC- Multiple Dose Cohorts
Time Frame: Baseline, Day 155
Population: The Pharmacodynamic Set included all participants who received at least 1 dose of study drug and had evaluable properdin concentration, CAP or complement classical pathway activity data. Here, Number of participants analyzed signifies those who were evaluable for this outcome measure. As per pre-specified analysis, only data for Cohorts 8 and 9 and the placebo arm were collected for this Outcome Measure.
Measure: Mean (Standard Deviation); unit: micrograms/milliliters
Arm/Group | Cohort 8: ALXN1820 150 mg SC (QW*5) | Cohort 9: ALXN1820 150 mg SC (QW*5) | All Placebo
Number analyzed (Participants) | 6 | 5 | 4
micrograms/milliliters | 6.018 (2.5094) | 9.878 (1.6731) | 0.418 (0.2806)

9. Secondary Outcome: Change From Baseline In Serum Concentrations of Free Properdin For ALXN1820 SC- Multiple Dose Cohorts
Time Frame: Baseline, Day 155
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: nanograms/milliliters
Arm/Group | Cohort 8: ALXN1820 150 mg SC (QW*5) | Cohort 9: ALXN1820 150 mg SC (QW*5) | All Placebo
Number analyzed (Participants) | 6 | 5 | 4
nanograms/milliliters | 3775.2 (1480.18) | 3762.0 (796.41) | 154.5 (480.34)

10. Secondary Outcome: Change From Baseline In Complement Alternative Pathway (CAP) Activity Using The Wieslab Alternative Pathway (AP) Assay For ALXN1820 SC And ALXN1820 IV-Single Dose Cohorts
Time Frame: Baseline, Day 127
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percentage of activity
Arm/Group | Cohort 1: ALXN1820 12.5 mg SC | Cohort 2: ALXN1820 50 mg SC | Cohort 3: ALXN1820 150 mg SC | Cohort 4: ALXN1820 450 mg SC | Cohort 5: ALXN1820 450 mg IV | Cohort 6: ALXN1820 1200 mg SC | Placebo
Number analyzed (Participants) | 5 | 6 | 5 | 4 | 5 | 6 | 11
percentage of activity | -15.6800 (19.06770) | 5.0833 (28.14281) | 1.6600 (18.75241) | 10.3750 (35.92282) | 3.100 (23.43683) | 6.6500 (20.32956) | 5.8091 (25.66349)

11. Secondary Outcome: Change From Baseline In Complement Alternative Pathway Activity Using The Wieslab Alternative Pathway Assay For ALXN1820 SC- Multiple Dose Cohorts
Time Frame: Baseline, Day 155
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: percentage of activity
Arm/Group | Cohort 8: ALXN1820 150 mg SC (QW*5) | Cohort 9: ALXN1820 150 mg SC (QW*5) | All Placebo
Number analyzed (Participants) | 7 | 6 | 4
percentage of activity | 27.9714 (34.63436) | 2.6667 (25.02420) | 7.0000 (15.05169)

12. Secondary Outcome: Number Of Participants With Positive Antidrug Antibodies (ADAs) To ALXN1820 SC And ALXN1820 IV
Time Frame: Baseline up to Day 155
Population: The Immunogenicity Set included all participants who had a predose and at least 1 postdose ADA sample collected. As per pre-specified analysis, only data for Cohorts 1-6, and Cohorts 8 and 9, and the placebo arm were collected for this Outcome Measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: ALXN1820 12.5 mg SC | Cohort 2: ALXN1820 50 mg SC | Cohort 3: ALXN1820 150 mg SC | Cohort 4: ALXN1820 450 mg SC | Cohort 5: ALXN1820 450 mg IV | Cohort 6: ALXN1820 1200 mg SC | Cohort 8: ALXN1820 150 mg SC (QW*5) | Cohort 9: ALXN1820 150 mg SC (QW*5) | All Placebo
Number analyzed (Participants) | 5 | 6 | 5 | 5 | 5 | 6 | 7 | 6 | 15
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0

13. Secondary Outcome: Absolute Bioavailability Of ALXN1820 SC
Description: The absolute bioavailability was expressed as ratio and was calculated as the geometric mean for the AUC[0-inf] for SC divided by the geometric mean for the AUC[0-inf] for IV. Least square means were calculated with cohort, treatment, and sequence as the fixed effects, and participant-participant (sequence) as a random effect.
Time Frame: Baseline up to Day 127
Population: The Pharmacokinetic Set included all participants who received at least 1 dose of study drug and had at least 1 post-dose PK concentration measured. Data for the arms reported is from the data collected based on pre-specified analysis.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Cohort 4: ALXN1820 450 mg SC
Number analyzed (Participants) | 5
Ratio | 89.307 [67.806 to 117.625]

ADVERSE EVENTS:
Time Frame: Baseline up to Day 155
Description: The Safety Set included all participants who received at least 1 dose of study drug.
Arm/Group | Cohort 1: ALXN1820 12.5 mg SC | Cohort 2: ALXN1820 50 mg SC | Cohort 3: ALXN1820 150 mg SC | Cohort 4: ALXN1820 450 mg SC | Cohort 5: ALXN1820 450 mg IV | Cohort 6: ALXN1820 1200 mg SC | Cohort 8: ALXN1820 150 mg SC (QW*5) | Cohort 9: ALXN1820 150 mg SC (QW*5) | All Placebo
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/6 | 0/5 | 0/5 | 0/5 | 0/6 | 0/7 | 0/6 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/6 | 0/5 | 0/5 | 0/5 | 0/6 | 0/7 | 0/6 | 0/15
Other Adverse Events (participants affected / at risk) | 4/5 | 6/6 | 2/5 | 4/5 | 4/5 | 6/6 | 6/7 | 5/6 | 11/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: ALXN1820 12.5 mg SC (N=5) | Cohort 2: ALXN1820 50 mg SC (N=6) | Cohort 3: ALXN1820 150 mg SC (N=5) | Cohort 4: ALXN1820 450 mg SC (N=5) | Cohort 5: ALXN1820 450 mg IV (N=5) | Cohort 6: ALXN1820 1200 mg SC (N=6) | Cohort 8: ALXN1820 150 mg SC (QW*5) (N=7) | Cohort 9: ALXN1820 150 mg SC (QW*5) (N=6) | All Placebo (N=15)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 3 (3) | 0 (0) | 2 (2)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 2 (3) | 0 (0) | 1 (2)
Upper respiratory tract infection (Infections and infestations) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinovirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatophytosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 4 (4)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 2 (3) | 1 (1) | 1 (2) | 0 (0) | 3 (4)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness exertional (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Migraine with aura (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tension headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Infusion site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heat exhaustion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post vaccination syndrome (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaccination complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intermenstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urine odour abnormal (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Immunisation reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-07-06): https://cdn.clinicaltrials.gov/large-docs/62/NCT04631562/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-28): https://cdn.clinicaltrials.gov/large-docs/62/NCT04631562/SAP_001.pdf